CLINICAL TRIAL: NCT01156324
Title: The Impact of an Online Stress Management Program on IVF Outcome
Brief Title: The Impact of an Online Stress Management Program on In Vitro Fertilization (IVF) Outcome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: Boston IVF (Other)
Responsible Party: Principal Investigator, Alice D. Domar, PhD, Alice D. Domar, PhD, Boston IVF
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100765
Record Dates: First submitted 2010-06-29; First posted 2010-07-02 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: IVF; Stress management
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Participants of the routine care control group will each receive a $50 gift certificate at the end of each IVF cycle for which they completed the questionnaires.
  Interventions: Behavioral: Online Stress Management Group (Upliv)
- Online Stress Management Group (Upliv) (Experimental): Personalized online stress management program consisting of weekly sessions which each include relaxation exercises, stress management strategies, and lifestyle modification advice. Participants in Upliv will also be given a set of personal care products as part of the program.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Online Stress Management Group (Upliv) — Personalized online stress management program
  Arms: Control
Behavioral: Control — Control group receiving routine care along with $50 gift certificate at end of cycle
  Arms: Online Stress Management Group (Upliv)

SUMMARY:
The goal of this study is to determine the impact of an online stress management program, which combines stress reduction and prevention strategies with personal care products/rituals which have relaxation properties, on pregnancy rates and psychological distress in women undergoing IVF for the first time.

DETAILED DESCRIPTION:
The relationship between stress and infertility has remained a subject of controversy for many years. Recent research indicates that stress has a strong negative impact on pregnancy rates in women undergoing in vitro fertilization (IVF). In addition, stress is the most common reason given by women who voluntarily terminate treatment.

In a recent study, women who participated in a group mind/body treatment program had higher pregnancy rates than control subjects. The impact of an online stress management program has never been studied in the infertile population. An online intervention would be far more accessible for many infertility patients.

ELIGIBILITY:
Inclusion Criteria:

* female Boston IVF patients
* day three FSH 12 or below
* day three estradiol 80 pg/ml or below
* able to read, understand and sign the informed consent in English
* using own eggs (not egg donor)
* willing and able to comply with study requirements
* must be well versed in using a personal computer and the internet and must have access to an internet-connected computer seven days per week

Exclusion Criteria:

* prescription antipsychotic medication
* previous diagnosis of borderline or narcissistic personality disorder
* previous or concurrent participation in a mind/body group

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rates | 1 year
  Clinical pregnancy rates will be recorded for IVF cycles 1 and 2.

SECONDARY OUTCOMES:
Psychological Status | 1 year
  Psychological status is assessed by the following scales: Perceived Stress Scale (PSS), State Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI), Social Readjustment Scale (SRS), Daily Monitoring Form (DMF). Other than the DMF, these are all published validated scales.

CONTACTS AND LOCATIONS:
Overall Officials: Alice D Domar, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No